CLINICAL TRIAL: NCT06733909
Title: Clinical Evaluation of Digital Versus Prefabricated Primary Crowns For Restoration of Pulpotomized Primary Molars: A Randomized Clinical Trial
Brief Title: Clinical Outcomes of Digital vs Prefab Crowns for Pulpotomized Primary Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-2
Record Dates: First submitted 2024-05-28; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-04

CONDITIONS: Pulpotomized Primary Molars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NuSmile Zirconia crowns (Active Comparator): Prefabricated pediatric Zirconia crowns offer an excellent alternative to full-coverage crowns when restoring deciduous teeth with a sizeable carious defect
  Interventions: Other: Restoration of Pulpotomized Primary Molars using NuSmile Zirconia crowns
- BioFlx crowns (Experimental): The Bioflex crown has been introduced in pediatric practice as a synthetic crown that will provide better adaptation, durability, and ease of handling with improved aesthetic properties compared to conventional crowns
  Interventions: Other: Restoration of Pulpotomized Primary Molars using BioFlx crowns
- Digital VITA ENAMIC crowns (Experimental): is a hybrid ceramic with a dual network structure that combines the best characteristics of ceramic and composite. Fast and efficient CAM fabrication; for minimally invasive reconstructions, tooth-like material properties.
  Interventions: Other: Restoration of Pulpotomized Primary Molars using Digital VITA ENAMIC crowns (CAD/CAM blanks)

INTERVENTIONS:
Other: Restoration of Pulpotomized Primary Molars using NuSmile Zirconia crowns — Prefabricated pediatric Zirconia crowns offer an excellent alternative to full-coverage crowns when restoring deciduous teeth with a sizeable carious defect. These crowns have high flexural strength, allowing them to resist crack propagation. The additional benefits of these crowns are the ability to replace metals due to extremely high strength and toughness, higher resistance to chemicals, and superior erosion resistance
  Arms: NuSmile Zirconia crowns
Other: Restoration of Pulpotomized Primary Molars using BioFlx crowns — The Bioflex crown has been introduced in pediatric practice as a synthetic crown that will provide better adaptation, durability, and ease of handling with improved aesthetic properties compared to conventional crowns. The Bioflex crown may provide a promising result in terms of the clinician's and parental satisfaction as aesthetic is a prime concern for parents and children in this era. The limitations of the studies on this type of crowns will require more studies with more detailed clinical observation and larger sample size to provide more rigorous results.
  Arms: BioFlx crowns
Other: Restoration of Pulpotomized Primary Molars using Digital VITA ENAMIC crowns (CAD/CAM blanks) — is a hybrid ceramic with a dual network structure that combines the best characteristics of ceramic and composite. Fast and efficient CAM fabrication; for minimally invasive reconstructions, tooth-like material properties.
  Arms: Digital VITA ENAMIC crowns

SUMMARY:
NuSmile Zirconia crowns: Prefabricated pediatric Zirconia crowns offer an excellent alternative to full-coverage crowns when restoring deciduous teeth with a sizeable carious defect. These crowns have high flexural strength, allowing them to resist crack propagation. The additional benefits of these crowns are the ability to replace metals due to extremely high strength and toughness, higher resistance to chemicals, and superior erosion resistance. Zirconia crowns are biocompatible, autoclavable, and equal to or more durable than natural enamel.

DETAILED DESCRIPTION:
Since the introduction of primary Zirconia crowns, several studies have reported their clinical success. Severely mutilated primary anterior teeth showed that NuSmile Zirconia crowns (NuSmile Ltd., Houston, TX, United States) offered superior esthetics and durability with remarkable gingival responses up to 24 months. A clinical study on the wear behavior of primary enamel against Zirconia crowns demonstrated the lowest wear rate of primary enamel. A retrospective study that evaluated the clinical success and parental satisfaction showed a considerable percentage (89%) of parents were highly satisfied by the crowns' size, color, and form.

BioFlx crowns: The Bioflex crown has been introduced in pediatric practice as a synthetic crown that will provide better adaptation, durability, and ease of handling with improved aesthetic properties compared to conventional crowns. The Bioflex crown may provide a promising result in terms of the clinician's and parental satisfaction as aesthetic is a prime concern for parents and children in this era. The limitations of the studies on this type of crowns will require more studies with more detailed clinical observation and larger sample size to provide more rigorous results. Digital VITA ENAMIC crowns (CAD/CAM blanks): is a hybrid ceramic with a dual network structure that combines the best characteristics of ceramic and composite. Fast and efficient CAM fabrication; for minimally invasive reconstructions, tooth-like material properties. Vita Enamic has an 9 elastic modulus of 30-32 GPa and resembles dental hard tissues, enabling it to mimic the biomechanical properties of natural teeth. Moreover, Vita Enamic has the advantage of preserving the antagonist teeth from abrasion and performing better at heavy occlusal stresses because it has the ability to resist crack initiation and progression. CAD/CAM technology is an innovative method of producing indirect restorations in primary teeth. With the help of the design software, the clinician can produce ideal occlusal and proximal contact points and a better marginal fit at the gingival wall. Moreover, it involves a shorter clinical working time which is beneficial for children's patients, less wear of the opposing dentition, and the choice of more biocompatible materials. However, there are limited cases of restorations on primary teeth with CAD/CAM technology Computer-aided design and manufacturing (CAD/CAM) technology have made enormous improvements since its introduction. Nowadays, this technology is available directly in dental clinics and it is capable, via its software, of fabricating (customized) full ceramic crowns, inlays, onlays, and veneers for permanent dentition at one appointment.

To date, most clinical studies of prefabricated crowns have been conducted on anterior teeth. There is a lack of information regarding the longevity of such crowns on primary teeth. Therefore, the objective of the present study was to evaluate the clinical success rate of NuSmile pediatric Zirconia, BioFlx crowns and Digital VITA ENAMIC crowns (CAD/CAM blanks) using 3 Shape TRIOS® Intraoral Scanner in primary posterior teeth up to one year.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 5 and 9 years old.
2. Positively cooperative children.
3. Children having a restorable pulpotomized primary tooth.
4. Primary molars with no spontaneous or provoked pain
5. Teeth to be included should be fully erupted, have functional occlusion.
6. The crowned molar is in contact with at least one adjacent molar medially with primary first molar and- or laterally with permanent first molar (standard for posterior crowns).

Exclusion Criteria:

1. Patients with systemic diseases (congenital or rheumatic heart disease, hepatitis, nephritis, tumor, cyclic neutropenia, leukemia, and children on long-term corticosteroid therapy).
2. Un-cooperative patients.
3. The child having oral parafunctional habits
4. Un-restorable primary molars (Grossly broken-down primary molars that have decay extending way under the gingiva and tooth with root caries).

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 12 months
  aesthetics, functional and biological criteria of the restorations

CONTACTS AND LOCATIONS:
Locations (1):
- MSA University, El-Sheikh Zayed City, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No